CLINICAL TRIAL: NCT01179035
Title: The Impact of Parolee-Targeted Care Versus Expedited Usual Care on Health Care Utilization and Recidivism
Brief Title: Evaluation of Transitions Clinic: A Post-Release Clinic for Recently Released Parolees With Chronic Medical Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Transitions Clinic (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Clemens Hong, MD/MPH, Transitions Clinic
Allocation: Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: Transitions001
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Health Services Research, Prisons, Delivery of Health Care, Vulnerable Populations, Community Health Aides
Keywords: Post-release, community health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expedited Primary Care (Active Comparator): Following randomization, subjects receive ongoing primary care in the San Francisco Department of Public Health affiliated primary care network. Appointments are expedited with safety-net primary care providers.
  Interventions: Other: Expedited Primary Care
- Transitions Clinic - Parolee Targeted Care (Experimental): Following randomization, subjects in this arm receive ongoing primary care in a parolee-targeted clinic. Parolee-targeted care includes care from clinicians with a knowledge of the impacts of incarceration on health and experience caring for formerly incarcerated patients, a community health worker that works in medical and social services coordination and chronic disease education, and linkages with community-based organizations serving formerly incarcerated individuals.
  Interventions: Other: Transitions Clinic - parolee-targeted care

INTERVENTIONS:
Other: Transitions Clinic - parolee-targeted care — Subjects receive ongoing primary care from the Transitions Clinic versus ongoing primary care in the San Francisco Department of Public Health affiliated primary care network.
  Arms: Transitions Clinic - Parolee Targeted Care
Other: Expedited Primary Care — Following randomization, subjects receive ongoing primary care in the San Francisco Department of Public Health affiliated primary care network. Appointments are expedited with safety-net primary care providers.
  Arms: Expedited Primary Care

SUMMARY:
The purpose of this study is to study the effectiveness of the Transitions Clinic, a post-release clinic for parolees with chronic medical conditions, in achieving increased primary care engagement, lower rates of inappropriate hospitalizations, psychiatric emergency service and emergency department use, and decreased recidivism.

We hypothesize that subjects receiving parolee-targeted care in the Transitions Clinic will have increased rates of non-emergency department ambulatory care and outpatient mental health care, lower rates of hospitalization, psychiatric emergency service (PES) utilization, emergency department (ED) utilization, decreased total hospital length of stay, and decreased recidivism compared to patients receiving primary care from other safety-net providers.

DETAILED DESCRIPTION:
With ever increasing numbers of released inmates, policymakers are developing policy initiatives and directing funding towards community reentry programs for recent parolees to decrease recidivism and improve health outcomes. These reentry programs are comprehensive efforts that coordinate social and medical services for recently incarcerated people to achieve these aims. Due to documented poor health outcomes in this population and the resultant costs on the public health system, provision of medical care will be an integral part of these reentry initiatives. The manner in which medical care is incorporated into community reentry programs and directed to recently released prisoners needs to be studied to guide architects of reentry programs, policymakers and allocation of funding.

The Transitions Clinic (TC) was founded to address the medical needs of recently released prisoners. The TC is a pilot project designed to target primary care medical services to parolees in San Francisco and aid in coordination of medical and social services. It operates within the San Francisco Department of Public Health(SFDPH)-affiliated Community Health Network (CHN) and is part of the Safe Communities Reentry Council, a city-wide, collaborative effort of the Sheriff's office, Public Defenders' office and local community organizations to improve reentry services and outcomes for the 1500 annual parolees to San Francisco.

The proposed project will prospectively examine the effectiveness of the TC in achieving increased primary care engagement, decreased acute health care utilization and decreased recidivism. After intake in the TC, patients will be randomized to continued, parolee-targeted care in TC versus referral to safety net medical providers for non-targeted care. We believe that the results of the study will assist policymakers by improving our understanding of the:

1. effect of targeted and non-targeted medical care provision to post-release prisoners on primary care engagement and utilization
2. effect of targeted and non-targeted medical care provision to post-release prisoners on inpatient hospitalizations and emergency room and psychiatric emergency service utilization.
3. effect of targeted and non-targeted care provision to post-release prisoners on recidivism
4. costs for provision of targeted versus non-targeted medical care to post-release prisoners (Do we want to do a cost analysis?)

ELIGIBILITY:
Inclusion Criteria:

* All adult parolees to San Francisco
* Must have one chronic condition or age >50 years old

Exclusion Criteria:

* Children
* Subjects who already have an established primary care provider in San Francisco

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)

PRIMARY OUTCOMES:
Acute Care Utilization | 6 months
  Hospitalization and hospital length of stay and psychiatric emergency and emergency department utilization

SECONDARY OUTCOMES:
Primary Care Engagement | 6 months
  Non-emergency department visits to ambulatory primary care and mental health providers
Recidivism | 6 months
  Rate of re-incarceration during study period

CONTACTS AND LOCATIONS:
Locations (1):
- Southeast Health Center, San Francisco, California, United States

REFERENCES:
- [Background] Wang EA, Hong CS, Samuels L, Shavit S, Sanders R, Kushel M. Transitions clinic: creating a community-based model of health care for recently released California prisoners. Public Health Rep. 2010 Mar-Apr;125(2):171-7. doi: 10.1177/003335491012500205. PMID 20297743